CLINICAL TRIAL: NCT05454904
Title: Design, Implementation, and Prospective Evaluation of a Mediterranean Diet- and Psychological Well-being Theory-based Intervention to Reverse Metabolic Syndrome, a Highly Prevalent Chronic Disease Risk Condition in Chile
Brief Title: Mediterranean Diet- and Psychological Well-being Theory-based Intervention to Reverse Metabolic Syndrome in Chile
Acronym: CHILEMED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 190606013; 1201607 (Other: FONDECYT - ANID - Chile)
Record Dates: First submitted 2020-09-12; First posted 2022-07-12 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-05

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Mediterranean diet; Psychological well-being
MeSH Terms: conditions — Metabolic Syndrome; Psychological Well-Being | interventions — Diet, Fat-Restricted; Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Three parallel-group randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low fat diet (Active Comparator): The low fat diet group will be counseled to consume a dietary pattern with fat restriction including food intake based in the pre-specified nutritional criteria.
  Interventions: Behavioral: Low fat diet
- Mediterranean diet alone (Active Comparator): The Mediterranean group will receive indications to consume a locally adapted and feasible dietary pattern including characteristic Mediterranean foods based on Chilean food availability.
  Interventions: Behavioral: Mediterranean diet
- Mediterranean diet plus psychological well-being support (Active Comparator): The Mediterranean diet + well-being intervention group will be subject to intake a locally adapted and feasible pattern of Mediterranean foods available in Chile in combination with a psychological well-being theory-based intervention.
  Interventions: Behavioral: Mediterranean diet; Behavioral: Mediterranean diet plus psychological well-being support

INTERVENTIONS:
Behavioral: Low fat diet — The low fat diet group will be counseled to consume a dietary pattern with fat restriction including food intake based in the following criteria: 1) <3 teaspoons/day of olive or Canola oil and <3 units/week of avocado, 2) removal of visible fat from meats before cooking or from cooked dishes before intake, 3) ≤1 serving per week fat-rich meats, hamburger, commercial ground meat, sausage, cured ham, bacon and salami, 4) daily consumption of low fat dairy products, 5) ≤1 serving/week of butter, margarine, lard, mayonnaise, milk cream, or milk- based ice cream, 6) ≤1 time/week intake of fatty fish or seafood, 7) ≤1 serving per week of commercial sweets or industrial bakery products (not homemade), and 8) ≤1 time/week consumption of nuts (including peanuts), potato chips, French fries, or commercial snacks. This intervention arm will be supplemented with powdered low fat milk (3 kgs/month) for daily use.
  Arms: Low fat diet
Behavioral: Mediterranean diet — The Mediterranean diet group will receive dietary recommendations as follows: 1) use of olive oil (>3 teaspoons/day), 2) Canola oil as second fat source for cooking and dressing or >3 units/week of avocado; 3) ≥3 daily servings of vegetables (at least one of them as fresh vegetables in a salad), 4) ≥2 daily servings of fresh fruits; 5) ≥2 weekly servings of legumes; 6) >2 weekly servings of fresh, canned or frozen fish (at least one serving of oily fish)/seafood; 7) ≥2 weekly servings of nuts/seeds; 8) 4-8 servings/week of white meats (poultry or turkey without skin) instead of 9) fatty or processed meats (<1 serving/week), 10) ≥2 daily servings of whole grains, 11) ≥1 daily/serving of low fat and fermented dairy products, 12) <1 daily/serving of whole fat dairy products, 13) ≤1 daily/serving of sugary snacks, drinks or juices and <4 teaspoons/daily of sugar, and 14) moderate (1-2 drinks/day) wine consumption with meals.
  Arms: Mediterranean diet alone; Mediterranean diet plus psychological well-being support
Behavioral: Mediterranean diet plus psychological well-being support — This group will be subjected to the same Mediterranean diet pattern indicated previously as well as to a psychological well-being intervention that will include a variety of components/activities, embracing values, purpose, self-acceptance, character strengths, emotional regulation, dealing with negativity, goal-setting, mindfulness, savoring, gratitude, autonomy, relationships, social interactions, and prosocial behavior.
  Arms: Mediterranean diet plus psychological well-being support

SUMMARY:
Promotion of MedDiet adherence and psychological well-being in Chile offers a great potential to confront our ongoing epidemiological transition to increased risk factors and non-communicable chronic diseases. The main aims of this clinical trial are to design, implement, and evaluate the impact of a MedDiet- and psychological well-being-based intervention on reversal rate of MetS -compared to a control low fat diet- in Chilean adult population.

DETAILED DESCRIPTION:
BACKGROUND: Non-communicable diseases (NCDs) are currently major causes of morbidity and mortality as well as economic healthcare burden worldwide, including Chile. Predisposing psychosocial as well as lifestyle risk factors -such as an unhealthy diet- have driven this global increase in NCDs. Overall, the ongoing epidemiological transition and current health situation in our country calls out for an urgent need to further evaluation of disease-related psychosocial factors and diet as well as definition of evidence-based feasible and effective nutritional interventions in the Chilean population. In addition, dietary interventions may be more easily incorporated and followed if provided and supported by theory-based and contextually grounded psychological approaches within a comprehensive positive psychosocial framework.

Currently, the Mediterranean diet (MedDiet) is one of the healthiest dietary patterns based on observational studies in developed countries showing that adherence to this food intake pattern associates with lower prevalence/incidence of several NCDs, including metabolic syndrome (MetS), and reduced total mortality. Far fewer interventional studies -essentially performed in Europe and some of them questioned due to methodological issues and others with inconsistent findings- have reported favorable effects of MedDiets on clinical outcomes. Thus, impact of MedDiet on high-risk conditions (i.e., MetS) and clinical end-points in populations outside the Mediterranean Basin remains unknown. Thus, additional interventional studies about this dietary pattern on disease outcomes in more diverse populations, including our country, are needed.

A Mediterranean lifestyle goes beyond mere food intake: it includes promotion of psychosocial resources, community life as well as cultural traditions. Indeed, Mediterranean lifestyle is a real way of life that integrally promotes physical, mental, and social well-being. However, psychological well-being (PWB) is much more than absence mental disorders. From a positive framework, PWB encompasses emotional/subjective well-being together with effective psychological functioning within a favorable social context and has been associated with healthy behaviors, positive health outcomes, and longevity. Promotion of PWB is in fact an emerging goal in healthcare, shifting the focus from treating/preventing mental disease to enhancing positive aspects of mental health. If PWB interventions are feasible and effective in boosting adherence to health behaviors, they may become a cost-effective tool to improve biomarker, functional and clinical outcomes related to NCDs.

Based in this latter broad and positive psychosocial paradigm, promotion of PWB may facilitate acquisition and routine practice of healthy lifestyles, such as MedDiet, decreasing risk of NCDs. However, to our knowledge, PWB theory-based interventions have not been tested as a new approach to increase MedDiet adherence. Based on the multi-construct model of this theory, which is consistent with a Mediterranean lifestyle, a comprehensive PWB intervention program may increase adherence to MedDiet and -in turn- enhance its impact on chronic disease risk conditions such as MetS.

Remarkably, Central Chile has a Mediterranean-like environment and food production comparable to those present in Mediterranean countries. Chilean culinary traditions also use ingredients and cooking techniques similar to Mediterranean cuisine. Thus, promotion of MedDiet adherence in Chile offers a great potential to confront our ongoing epidemiological transition to increased risk factors and NCDs. Despite our geography, food production, culinary traditions, and potential health benefits, very few studies have evaluated the potential impact of MedDiet patterns on health and/or disease in Chilean subjects. Furthermore, these studies exhibit important methodological limitations, such as only cross sectional observational analysis or small sample sizes, no control comparators for interventions, lack of theory-based behavior change advice, and use of intermediate biomarkers rather than clinical end-points. Better designed intervention studies using a locally tailored MedDiet index, feasible dietary prescription, novel PWB advice strategies as well as comprehensive outcome evaluation are required to further support and more extensively implement this dietary pattern and its associated positive psychosocial features for NCD prevention and treatment in our population.

GUIDING HYPOTHESES. A psychological well-being theory-based behavioral support increases long-term MedDiet adherence and this nutritional intervention combined with promotion of psychological well-being is more effective at reversing MetS in Chilean subjects (primary outcome) and improving additional relevant biomarkers, clinical conditions, and well-being (secondary outcomes) compared to individuals following a low fat dietary pattern alone.

OVERALL AIMS: 1. To design a PWB intervention as well as to refine a MedDiet pattern adapted and contextualized to Chilean subjects; 2. To determine if a customized psychological well-being intervention facilitates initiation and long-term adherence to a MedDiet dietary pattern in Chilean subjects with MetS; 3. To demonstrate that a locally adapted MedDiet pattern in association with a psychological well-being intervention -versus a low fat diet alone- increases the reversal rate of MetS; and 4. To establish whether this dietary approach with or without a psychological intervention improves traditional and novel disease biomarkers as well as non-alcoholic fatty liver disease and psychological well-being -compared to a control low fat diet- in Chilean subjects with MetS.

METHODOLOGY. Overall, this proposal will design and implement a PWB theory-based behavior change strategy to increase MedDiet adherence and perform a clinical MedDiet intervention as main experimental research approaches. A tailored contextualized PWB intervention will be designed using information derived from focus group-based qualitative research. Then, a parallel-group randomized controlled clinical trial will be developed to determine the impact of MedDiet- and psychological well-being theory-based nutritional intervention on MetS (primary end-point), disease-associated biomarkers, fatty liver disease, depression, quality of life, and psychological well-being (secondary outcomes). Appropriate study protocols, anthropometric, questionnaire-based, biochemical, imaging, and clinical follow-up evaluations as well as proper statistical approaches will be implemented and applied in the RCT study.

SIGNIFICANCE AND IMPLICATIONS: If the main findings turn out as expected (psychological well-being intervention facilitates adherence to MedDiet and this combined intervention reduces MetS and improves related-secondary clinical and psychosocial outcomes), this research proposal will provide further evidence on the beneficial health effects of the MedDiet beyond the Mediterranean basin, particularly in our country. Based on this locally generated evidence, MedDiet associated with promotion of positive psychosocial resources may be more compellingly applied to promote physical health and well-being as well as to prevent and treat NCD at individual and population levels in Chile.

ELIGIBILITY:
Inclusion Criteria:

Adult men or women 25-70 years-old with existing metabolic syndrome defined as the presence of at least three of the following criteria: (i) abdominal obesity (waist circumference >90 cm in men or >80 cm in women), (ii) low HDL-cholesterol (<40 mg/dl in men or <50 mg/dl in women) or under HDL increasing drugs, (iii) high triglycerides (TG) (≥ 150 mg/dl) or under TG lowering drugs, (iv) high blood hypertension (blood pressure ≥ 130/85 mmHg) or under treatment, and (v) high blood glucose (fasting plasma glucose concentration ≥ 100 mg/dl) or under treatment.

Exclusion Criteria:

* Absence of written informed consent
* Inability/low chance of adherence to diets or attend scheduled visits
* Allergy or intolerance to foods included in either interventional diets
* Recent (<12 months) participation in weight loss program
* Obesity with BMI >35 kg/m2 or due to endocrine diseases, with exception of treated hypothyroidism
* Type 1 diabetes, unstable type 2 diabetes
* Uncontrolled high blood pressure
* Previous clinical atherosclerotic cardiovascular disease
* Use of medications such as weight loss drugs, oral corticoids, immunosuppressants or cytotoxic agents
* Advanced chronic liver disease
* Previous organ transplantation
* History of HIV-positive status or AIDS
* History of inflammatory bowel disease or major gastrointestinal surgery (bariatric surgery, bowel resection)
* Active psychiatric conditions: eating disorders, severe depression, bipolar disorder, schizophrenia
* Short (<2 years) life expectancy
* Current or previous (within the last year) participation in other clinical trials with dietary or drug interventions
* Institutionalized subjects
* Additional conditions that may limit adherence to the study

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic syndrome | Month 12
  Metabolic syndrome is diagnosed when three out of five criteria from the NCEP ATPIII definition are present. The nutritional interventions will determine metabolic syndrome reversal when participants exhibit from 0 to 2 diagnostic criteria at the end of the study.

SECONDARY OUTCOMES:
Mediterranean Dietary adherence | Month 6 and 12
  Diet adherence to this food intake pattern will be assessed by the Chilean Mediterranean dietary index. Change in adherence to this diet will be evaluated as modification in the score (ranging from 0 to 14 points) during the interventions. Higher scores mean a better outcome.
Insulin Resistance | Month 6 and 12
  Insulin resistance will be assessed through the HOMA-IR index obtained by measuring fasting glucose (mg/dL) and fasting insulin (uU/mL).
Glucose homeostasis | Month 6 and 12
  Overall glucose homeostasis will be evaluated by measuring glycated hemoglobin (HbA1c)
Lipid profile | Month 6 and 12
  Fasting triglycerides, total cholesterol, and HDL-cholesterol (all expressed as mg/dL) will be assessed to categorize lipid changes.
High sensitivity C-reactive protein | Month 6 and 12
  High sensitivity C-reactive protein will be determined as pro-inflammatory and prognostic biomarker.
Plasma antioxidant capacity | Month 6 and 12
  Ferric reducing ability of plasma (FRAP) in fasting plasma samples of participants will be used to assess total plasma antioxidant activity.
Lipid peroxidation | Month 6 and 12
  Oxidized low-density lipoprotein (oxLDL) will be measured as lipid peroxidation biomarker
Serum protein oxidation | Month 6 and 12
  Advanced oxidation protein products (AOPP) will be measured in serum samples as a biomarker of oxidative stress in proteins.
Body mass index (BMI) | Month 6 and 12
  BMI will be calculated using weight and height in order to define the nutritional status of the patients
Abdominal obesity | Month 6 and 12
  Abdominal/central obesity will be evaluated by measuring waist circumference
Blood pressure control | Month 6 and 12
  Systolic/diastolic blood pressures will be assessed.
Type 2 diabetes mellitus | Month 6 and 12
  Type 2 diabetes mellitus will be assessed based on ADA definitions, including fasting glycemia ≥ 126 mg/dl, 2-h glycemia ≥ 200 mg/dl after glucose challenge, HbA1C ≥6.5%, or patient with hyperglycemic symptoms and random glycemia ≥ 200 mg/dl.
Psychological well-being | Month 6 and 12
  The Ryff's multidimensional questionnaire/scale will be used to assess psychological well-being levels. Change in well-being will be evaluated as modification in the overall scale score (from 29 to 174 points) during the interventions. Higher scores means a better psychological well-being outcome.
Positive mental health | Month 6 and 12
  Mental Health Continuum-short form questionnaire will be applied to assess positive emotional, psychological, and social well-being
Emotional affectivity | Month 6 and 12
  Positive and Negative Affect Schedule survey will evaluate emotional affectivity
Life, quality of | Month 6 and 12
  Quality of life will be assessed using the health-related quality of life (HRQoL) multidimensional SF-36 questionnaire. This questionnaire evaluates 8 dimensions using specific scales, each one ranging from 0 to 100 points. Higher scores indicate better quality of life.
Psychological illness | Month 6 and 12
  Psychological illness will be assessed using the DASS-21 self-reported questionnaire. This questionnaire includes depression, anxiety and stress scales, each one ranging from 0 to 21 points. Higher scores indicate worse psychological illness.

CONTACTS AND LOCATIONS:
Overall Officials: Attilio Rigotti, Principal Investigator — Professor
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dussaillant C, Echeverria G, Urquiaga I, Velasco N, Rigotti A. [Current evidence on health benefits of the mediterranean diet]. Rev Med Chil. 2016 Aug;144(8):1044-1052. doi: 10.4067/S0034-98872016000800012. Spanish. PMID 27905651
- [Background] Echeverria G, Urquiaga I, Concha MJ, Dussaillant C, Villarroel L, Velasco N, Leighton F, Rigotti A. [Validation of self-applicable questionnaire for a Mediterranean dietary index in Chile]. Rev Med Chil. 2016 Dec;144(12):1531-1543. doi: 10.4067/S0034-98872016001200004. Spanish. PMID 28393987
- [Background] Urquiaga I, Echeverria G, Dussaillant C, Rigotti A. [Origin, components and mechanisms of action of the Mediterranean diet]. Rev Med Chil. 2017 Jan;145(1):85-95. doi: 10.4067/S0034-98872017000100012. Spanish. PMID 28393974
- [Background] Echeverria G, McGee EE, Urquiaga I, Jimenez P, D'Acuna S, Villarroel L, Velasco N, Leighton F, Rigotti A. Inverse Associations between a Locally Validated Mediterranean Diet Index, Overweight/Obesity, and Metabolic Syndrome in Chilean Adults. Nutrients. 2017 Aug 11;9(8):862. doi: 10.3390/nu9080862. PMID 28800091
- [Background] Echeverria G, Dussaillant C, McGee EE, Mena C, Nitsche MP, Urquiaga I, Bitran M, Pedrals N, Rigotti A. Promoting and Implementing the Mediterranean Diet in the Southern Hemisphere: the Chilean Experience. Eur J Clin Nutr. 2019 Jul;72(Suppl 1):38-46. doi: 10.1038/s41430-018-0307-7. PMID 30487560
- [Background] Echeverria G, Tiboni O, Berkowitz L, Pinto V, Samith B, von Schultzendorff A, Pedrals N, Bitran M, Ruini C, Ryff CD, Del Rio D, Rigotti A. Mediterranean Lifestyle to Promote Physical, Mental, and Environmental Health: The Case of Chile. Int J Environ Res Public Health. 2020 Nov 16;17(22):8482. doi: 10.3390/ijerph17228482. PMID 33207718
- [Background] Figueroa C, Echeverria G, Villarreal G, Martinez X, Ferreccio C, Rigotti A. Introducing Plant-Based Mediterranean Diet as a Lifestyle Medicine Approach in Latin America: Opportunities Within the Chilean Context. Front Nutr. 2021 Jun 25;8:680452. doi: 10.3389/fnut.2021.680452. eCollection 2021. PMID 34249989